CLINICAL TRIAL: NCT07167940
Title: RAPID5: Rapid Acceleration Process for Intensive Treatment of PTSD in 5 Days
Brief Title: Rapid Acceleration Process for Intensive Treatment of PTSD in 5 Days
Acronym: RAPID5
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHBP-001-25S; 1I01RD001578-01A2 (Other Grant/Funding Number: VHA ORD CSRD)
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: PTSD
Keywords: Post-traumatic Stress Disorder; Transcranial Magnetic Stimulation; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TMS (Active Comparator): Active transcranial magnetic stimulation
  Interventions: Device: Transcranial magnetic stimulation
- Sham TMS (Sham Comparator): Non-active/sham transcranial magnetic stimulation
  Interventions: Device: Sham transcranial magnetic stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — iTBS; 50 Hz triplets given at 5 Hz frequency with a cycle time of 2 seconds on and 8 seconds off). There will be 60 cycles for a total of 1800 pulses
  Other Names: TMS
  Arms: Active TMS
Device: Sham transcranial magnetic stimulation — Sham iTBS; 50 Hz triplets given at 5 Hz frequency with a cycle time of 2 seconds on and 8 seconds off). There will be 60 cycles for a total of 1800 pulses
  Other Names: Sham TMS
  Arms: Sham TMS

SUMMARY:
Veterans with posttraumatic stress disorder (PTSD) need more effective treatments. Existing options can have limited adherence and can be very time-consuming. As such, alternative interventions are needed. Transcranial magnetic stimulation (TMS) has been FDA-cleared for depression since 2008 and has recently been cleared to treat smoking cessation and obsessive-compulsive disorder. It has demonstrated promise for reducing PTSD symptom severity but standard TMS has a significant time requirement. This study will compare an accelerated 5-day form of TMS versus sham for PTSD, characterizing efficacy and durability. This project will provide important information that can be implemented in the near term for Veterans with PTSD.

DETAILED DESCRIPTION:
The primary research question of the proposed study is: Can transcranial magnetic stimulation (TMS) effectively treat posttraumatic stress disorder in Veterans using a pragmatic accelerated approach? The investigators address the need to improve symptom severity in this population utilizing the RAPID5 TMS protocol which delivers five treatments per day over the course of five days. The proposed four-year randomized controlled trial will compare the RAPID5 protocol to a Sham TMS Control Condition. The primary aim of the proposed research is to evaluate the efficacy of TMS to ameliorate PTSD symptoms in Veterans. The second aim is to examine the durability of PTSD symptom reduction resultant from the RAPID5 protocol. Given the high rate of mild traumatic brain injury (mTBI) among Veterans with PTSD, the exploratory aims of the proposed research seek to assess the contribution of mTBI in the context of PTSD on TMS outcomes.

Exploratory aims of the proposed research are: 1) examine whether mTBI status moderates PTSD symptom reduction, 2) assess whether differences in executive functioning moderate or mediate PTSD symptom reduction in Veterans with and without mTBI, and 3) will RAPID5 result in improved executive functioning in Veterans with PTSD.

These aims will be testing in a double-blind randomized controlled trial which will compare the efficacy of RAPID5 to sham TMS. This trial will include 90 Veterans meeting criteria for PTSD ages 18-70 with half randomized to RAPID5 and half randomized to sham TMS. For the RAPID5 condition, Veterans will receive five treatments per day for five consecutive business days. This protocol is based on evidence from previous work in depression and pilot data collected within the national Clinical TMS Program. Veterans randomized to the sham control condition will receive five treatments per day for five consecutive business days. After completion of the active treatment phase, Veterans will be assessed at two follow-up timepoints: 1 month and 3 months posttreatment.

Participants will complete several assessments, including but not limited to semi-structured clinical interviews, symptom self-report rating measures, quality of life measures, and neuropsychological measures assessing executive functioning. The goal is to provide evidence of the efficacy of an accelerated TMS treatment protocol in reducing PTSD symptom severity, resulting in an easily implementable VA healthcare systemwide implementation of this protocol across the VA enterprise.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic PTSD, meeting DSM-5 criteria.
* Eligible Veterans (regardless of sex) will be between the ages of 18-70.
* Symptomatic despite ongoing stable treatment (medications, psychotherapy, etc.) for at least 6 weeks before study procedures.
* Ongoing medications and psychotherapy will be allowed to continue unchanged during the study.
* For safety, participants must meet established screening criteria for magnetic resonance imaging (MRI). This is implemented as a conservative measure given the novel application of TBS in this population since MRI involves magnetic fields at a similar intensity to those emitted from the stimulation coil. These measures require a patient not to have the following (unless MRI-safe): A cardiac pacemaker, implanted device (deep brain stimulation) or metal in the brain, cervical spinal cord, or upper thoracic spinal cord.
* Willingness to participate in a clinical trial for approximately 4 to 6 months (consisting of a treatment phase with a 4-month follow-up period).
* Veterans must also be willing and able to comply with all study-related procedures and visits and be capable of independently reading and understanding information materials and providing written informed consent.
* Sufficient visual and auditory acuity to allow neuropsychological testing.

Exclusion Criteria:

Psychiatric Exclusions

* Primary psychotic disorder, bipolar I disorder, and greater than moderate substance use disorder (within the last month, excluding nicotine/caffeine, assessed by a urine drug screen as indicated), determined by the Mini International Neuropsychiatric Interview (MINI).
* Active suicidal intent or plan, as detected on screening instruments or in the investigator team's opinion, is likely to attempt suicide within 6 months.
* The presence of any other condition or circumstance that, in the opinion of the investigator team, has the potential to prevent study completion and/or to have a confounding effect on outcome assessments.

Medical Exclusions

* History of neurological disorder (e.g., multiple sclerosis, seizure disorder, etc.) or systemic illness affecting CNS function (e.g., liver failure, kidney failure, congestive heart failure, metastatic cancer) or that could meaningfully impact cortical excitability.
* Acute illness or unstable chronic illness, e.g., history of severe liver disease (cirrhosis, esophageal varices, ascites, portal hypertension, hepatic encephalopathy).
* Pregnant or breastfeeding and planning to become pregnant within the next 3 months.
* Have a mass lesion, cerebral infarct, or other neuroanatomical abnormality located at the TMS treatment site (DLPFC); a lifetime history of a) seizure disorder b) primary or secondary CNS tumors c) stroke or d) cerebral aneurysm.
* Greater than mild traumatic brain injury (following VA/DoD definitions).
* Inability to read, unable to verbalize understanding, and voluntarily sign the Informed Consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-03-09 (Estimated); Primary Completion 2030-01-09 (Estimated); Study Completion 2030-02-02 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for the DSM-5 | T1:Baseline, T2: Post-Treatment, T3: One month post treatment, & T4: 3 months post-treatment
  Measure of the number and severity of PTSD symptoms. A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items. Higher scores indicate more severe PTSD.

SECONDARY OUTCOMES:
Executive Functioning | T1: Baseline, T2: Post-Treatment, & T4 3 months post treatment
  A set of several neuropsychological measures used to assess executive functioning skills. Administered measures will be transformed into standard scores in order to compare across various measures and create an overall aggregate score. Range will be -2.50 to 2.50 where higher scores indicate better functioning.
Pittsburgh Sleep Quality Index | T1:Baseline, T2: Post-Treatment, T3: One month post treatment, & T4: 3 months post-treatment
  Measure of sleep disturbance and sleep quality. Adding up the average scores of the seven factors gives a global PSQI score from 0 to 21, with where lower scores denote a healthier sleep quality.
Short-Form-36 | T1:Baseline, T2: Post-Treatment, T3: One month post treatment, & T4: 3 months post-treatment
  Measure of quality of life consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability

CONTACTS AND LOCATIONS:
Overall Officials: Michelle R Madore, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (2):
- United States (2):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No